CLINICAL TRIAL: NCT06873009
Title: Cognitive Behavioural Therapy for Smoking Cessation in Incarcerated Men: Efficacy and Predictors of Treatment Outcomes
Brief Title: Can Cognitive Behavioural Therapy Help Incarcerated Men Quit Smoking? Efficacy and Predictors of Treatment Outcomes
Acronym: PriSanTabac
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Collaborators: Paris Nanterre University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24.05937.000428
Record Dates: First submitted 2025-03-07; First posted 2025-03-12 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-02

CONDITIONS: Tobacco Use; Smoking Cessation; Cognitive Behavioral Therapy; Prisoners
Keywords: Tobacco use; Smoking cessation; Cognitive Behavioral Therapy; Prisoners
MeSH Terms: conditions — Tobacco Use; Smoking Cessation | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: This study is a three-arm randomized controlled trial (RCT) with a parallel design. Participants are randomly assigned to one of three groups: a cognitive-behavioral therapy (CBT) intervention, a health education program, or a waitlist control group. The study aims to evaluate the efficacy of the CBT intervention in helping incarcerated individuals quit smoking, compared to a health education program and a waitlist control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cognitive-Behavioral Therapy (CBT) group (Experimental): Participants in this group will receive a cognitive-behavioral therapy (CBT)-based intervention designed to help them quit smoking. The intervention consists of three structured group sessions (1.5 hours each) over three weeks, incorporating cognitive-behavioral, motivational, and emotional strategies.
  The sessions focus on:
  * Increasing motivation to quit smoking,
  * Managing cravings and withdrawal symptoms,
  * Developing coping strategies for stress,
  * Preventing relapse through behavioral and cognitive techniques. This program is adapted from Richmond et al. (2013) The program is based on Richmond et al. (2013) and has been further adapted for the specific context of this study and to align with current recommendations.
  Interventions: Behavioral: Cognitive-Behavioral Therapy (CBT) for Smoking Cessation
- Health Education Group (Active Comparator): Participants in this group will receive a single-session health education program (1 hour) focused on the risks of smoking and the mechanisms of tobacco addiction. The session is conducted in a group format by a psychologist-nurse team and aims to provide participants with knowledge about the effects of smoking on health.
  Interventions: Other: Health Education Session on Tobacco Use
- Waitlist Control Group (No Intervention): Participants in this group will not receive any intervention during the 3-month study period. They will be placed on a waitlist and will have the opportunity to participate in one of the two interventions (CBT or Health Education or both) after the study follow-up is completed.

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy (CBT) for Smoking Cessation — A structured three-session group intervention (1.5 hours per session over three weeks) using cognitive-behavioral and motivational strategies to enhance motivation, manage cravings, and prevent relapse.
  Associated Arm: CBT Group
  Arms: Cognitive-Behavioral Therapy (CBT) group
Other: Health Education Session on Tobacco Use — A single-session group intervention (1 hour) providing information on the health risks of tobacco use, addiction mechanisms, and the long-term benefits of quitting smoking.
  Associated Arm: Health Education Group
  Arms: Health Education Group

SUMMARY:
The goal of this clinical trial is to evaluate whether a brief group-based psychological intervention using cognitive-behavioral therapy (CBT) helps people in prison quit smoking. Researchers will compare this intervention to a health education program and a control group (waitlist) to see which approach is most effective.

The main questions this study aims to answer are:

* Does the CBT-based group intervention help more participants quit smoking compared to the health education group and the control group?
* Do participants in the CBT-based group intervention smoke fewer cigarettes per day one month after the intervention compared to the other groups?
* Do participants in the CBT-based group intervention have lower nicotine dependence ?
* What individual factors (e.g., motivation to quit, nicotine dependence, craving intensity, self-efficacy, withdrawal symptoms, anxiety, depression, ADHD, and PTSD) predict success in the CBT and Health education groups?

Participants will be randomly assigned to one of three groups:

* CBT group: Three group sessions (1.5 hours each) using CBT and motivational approaches to quitting smoking.
* Health education group: One group session (1 hour) providing information on smoking and its health risks.
* Control group: No intervention for three months (waitlist). All participants will complete an initial assessment, attend their assigned group sessions, and return for follow-up visits at 1 month and 3 months. Their smoking status will be measured through self-reports and carbon monoxide (CO) expired levels.

ELIGIBILITY:
Inclusion Criteria:

* Male individuals currently incarcerated at Maison d'Arrêt Paris-La Santé.
* Aged 18 years or older at the time of inclusion.
* Current smoker, defined as having smoked daily in the past 30 days, or having an occasional smoking pattern of at least 5 cigarettes during the past 30 days.
* Able to speak and understand French well enough to follow the study procedures and actively participate in group sessions.
* Sentence length of at least 6 months, or if in pretrial detention, having a scheduled trial date within at least 6 months.

Exclusion Criteria:

* Age under 18 years at the time of inclusion.
* Inability to speak and understand French well enough to follow the study procedures and actively participate in group sessions.
* Sentence length of less than 6 months, or if in pretrial detention, having a scheduled trial date in less than 6 months or no available information about the trial date.
* Severe cognitive impairment that affects comprehension and participation in the study.
* Unstable psychiatric conditions (including acute psychotic disorders, severe mood disorders, severe anxiety disorders).
* Individuals under legal guardianship or conservatorship (e.g., placed under tutelage, curatorship, or temporary guardianship).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Smoking Abstinence Verified by Carbon Monoxide (CO) Measurement at 1-Month Follow-Up | baseline to 1-month follow-up
  Smoking abstinence will be assessed through self-reported smoking status and verified by exhaled carbon monoxide (CO) levels measured using a CO monitor. Participants who self-report smoking abstinence and have a CO level below 8 parts per million (ppm) will be classified as abstinent. A CO level ≥8 ppm will indicate continued smoking.
Smoking Abstinence Verified by Carbon Monoxide (CO) Measurement at 3-Month Follow-Up | baseline to 3-month follow-up
  Smoking abstinence will be assessed through self-reported smoking status and verified by exhaled carbon monoxide (CO) levels measured using a CO monitor. Participants who self-report smoking abstinence and have a CO level below 8 parts per million (ppm) will be classified as abstinent. A CO level ≥8 ppm will indicate continued smoking.

SECONDARY OUTCOMES:
Number of Cigarettes Smoked Per Day at 1-Month Follow-Up | Baseline to 1-month follow-up
  The average number of cigarettes smoked per day, as self-reported by participants, will be assessed to evaluate changes in tobacco use. This outcome will be compared to baseline and between treatment groups (CBT, health education, control) at 1-month follow-up.
Number of Cigarettes Smoked Per Day at 3-Month Follow-Up | Baseline to 3-month follow-up
  The average number of cigarettes smoked per day, as self-reported by participants, will be assessed to evaluate changes in tobacco use. This outcome will be compared to baseline and between treatment groups (CBT, health education, control) at 3-month follow-up.
Nicotine Dependence (FTND Score) at 1-Month Follow-Up | Baseline to 1-month follow-up
  Nicotine dependence will be assessed using the Fagerström Test for Nicotine Dependence (FTND), with scores ranging from 0 (no dependence) to 10 (high dependence). Changes in scores will be compared from baseline to follow-up assessments and between treatment groups (CBT, health education, control).
Nicotine Dependence (FTND Score) at 3-Month Follow-Up | Baseline to 3-month follow-up
  Nicotine dependence will be assessed using the Fagerström Test for Nicotine Dependence (FTND), with scores ranging from 0 (no dependence) to 10 (high dependence). Changes in scores will be compared from baseline to follow-up assessments and between treatment groups (CBT, health education, control).
Smoking Craving (FTCQ-12 Score) at 1-Month Follow-Up | Baseline to 1-month follow-up
  Craving levels will be assessed using the French Tobacco Craving Questionnaire - 12 items (FTCQ-12), with total scores ranging from 12 (lowest craving) to 60 (highest craving). Changes in scores will be compared from baseline to follow-up assessments and between treatment groups (CBT, health education, control).
Smoking Craving (FTCQ-12 Score) at 3-Month Follow-Up | Baseline to 3-month follow-up
  Craving levels will be assessed using the French Tobacco Craving Questionnaire - 12 items (FTCQ-12), with total scores ranging from 12 (lowest craving) to 60 (highest craving). Changes in scores will be compared from baseline to follow-up assessments and between treatment groups (CBT, health education, control).
Self-Efficacy for Smoking Cessation at 1-Month Follow-Up | Baseline to 1-month follow-up
  Self-efficacy will be assessed using a Visual Analog Scale (VAS) ranging from 0 (not confident at all) to 10 (very confident). Changes in self-efficacy scores will be compared from baseline to follow-up assessments and between treatment groups (CBT, health education, control).
Self-Efficacy for Smoking Cessation at 3-Month Follow-Up | Baseline to 3-month follow-up
  Self-efficacy will be assessed using a Visual Analog Scale (VAS) ranging from 0 (not confident at all) to 10 (very confident). Changes in self-efficacy scores will be compared from baseline to follow-up assessments and between treatment groups (CBT, health education, control).
Predictors of smoking abstinence at 1-month follow-up | Baseline to 1 month follow-up
  Logistic regression will be used to examine predictors of abstinence (defined as self-reported 7-day abstinence confirmed by CO ≤ 8 ppm) at 1-month follow-up. Candidate predictors include baseline impulsivity (UPPS), anxiety and depression (HADS), nicotine dependence (FTND), education level, self-efficacy (VAS), motivation (ASSIST), ADHD symptoms (ASRS), PTSD symptoms (PCL-5), other substance use (ASSIST), and withdrawal symptoms (MNWS).
Predictors of smoking abstinence at 3-month follow-up | Baseline to 3 month follow-up
  Logistic regression will be used to examine predictors of abstinence (defined as self-reported 7-day abstinence confirmed by CO ≤ 8 ppm) at 3-month follow-up. Candidate predictors include baseline impulsivity (UPPS), anxiety and depression (HADS), nicotine dependence (FTND), education level, self-efficacy (VAS), motivation (ASSIST), ADHD symptoms (ASRS), PTSD symptoms (PCL-5), other substance use (ASSIST), and withdrawal symptoms (MNWS).

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Laqueille, MD, Head of Department, Principal Investigator — GHU Paris Psychiatrie et Neurosciences
Locations (1):
- Centre pénitentiaire Paris-La Santé (Paris-La Santé prison), Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No
Investigators do not plan to share individual participant data (IPD) for this study. The protocol submitted to the Ethics Committee (CPP) does not include any specific provision regarding data sharing, and participants were neither informed nor consented to such use. In accordance with ethical and regulatory requirements, as well as principles of confidentiality and data protection, investigators are therefore unable to make these data available to other researchers.

REFERENCES:
- [Background] Richmond R, Indig D, Butler T, Wilhelm K, Archer V, Wodak A. A randomized controlled trial of a smoking cessation intervention conducted among prisoners. Addiction. 2013 May;108(5):966-74. doi: 10.1111/add.12084. Epub 2013 Mar 11. PMID 23228222